CLINICAL TRIAL: NCT02401841
Title: Resolution of Neuro-muscular Block in Great Obese Patients: Neostigmine vs Sugammadex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: Policlinico 12
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Resolution of Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sugammadex: Patients treated with Sugammadex
  Interventions: Drug: Two different types of drug for resolution of neuro-muscular blockade
- Neostigmine: Patients treated with Neostigmine
  Interventions: Drug: Two different types of drug for resolution of neuro-muscular blockade

INTERVENTIONS:
Drug: Two different types of drug for resolution of neuro-muscular blockade

SUMMARY:
It is a observational prospective study. The aim of this study is to compare neostigmine vs sugammadex in the resolution of neuro-muscular blockade in great obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Great obese
* Videolaparoscopic surgery

Exclusion Criteria:

* Age under 18
* No acceptation of informed consent
* New York Heart Association > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Great obese patients undergoing videolaparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Differences in neuro-muscular block resolution time between two groups | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCC Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy